CLINICAL TRIAL: NCT05660096
Title: Validation of Cionic Neural Sleeve for Use in Pediatric Patients With Cerebral Palsy
Brief Title: Pediatric Neural Sleeve Validation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to obtain neural sleeve through partner company
Sponsor: University of California, Los Angeles (Other)
Collaborators: Cionic, Inc. (Industry)
Responsible Party: Principal Investigator, Rachel Thompson, MD, William and Patricia Oppenheim Presidential Chair in Pediatric Orthopaedics and Assistant Professor-in-Residence, UCLA Department of Orthopaedic Surgery, University of California, Los Angeles
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB#22-000971
Record Dates: First submitted 2022-11-28; First posted 2022-12-21 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Cerebral palsy patients will undergo gait analysis without the sleeve in the first phase of the study. The same patients will then under gait analysis with the sleeve in the second phase of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Patient with Cerebral Palsy, no intervention (No Intervention): Gait analysis of cerebral palsy patients without any intervention.
- Patient with Cerebral Palsy, with sleeve (Active Comparator): Gait analysis of cerebral palsy patients while wearing neural sleeve.
  Interventions: Device: Cionic Neural Sleeve NS-100

INTERVENTIONS:
Device: Cionic Neural Sleeve NS-100 — Sleeve applies neuromuscular stimulation as patients walk to help contract appropriate muscles at appropriate times.
  Other Names: External functional neuromuscular stimulator
  Arms: Patient with Cerebral Palsy, with sleeve

SUMMARY:
In individuals with cerebral palsy (CP), signals from the brain to the muscles that are required for coordinated walking are either poorly controlled or absent. This results in abnormal walking (or gait) patterns and difficulty with independent movement. The purposes of this study is to test a device - a wearable leg sleeve - that can measure the abnormal signals sent from the brain to the muscles and the resulting movements and then send signals to the muscles to help make walking easier and smoother.

20 participants with, and 10 participants without, CP are being asked to come to test the device at the Kameron Gait and Motion Analysis Center. This requires one visit, which will last approximately 2-4 hours. During this visit, participants will undergo a physical exam and will be fit for the device on their leg. The participant will be asked to move their legs while the device is on to calibrate the device, and then the participants will walk while the device is interpreting their movement patterns. Participants with cerebral palsy will additionally walk with the device on their leg in a "corrective mode," where the device will provide stimulation to certain muscles in their leg in order to improve the patient's walking pattern.

Last, participants will complete an instrumented gait analysis. Gait analysis involves recording movement patterns during walking using small reflective markers and sensor taped to the participant's legs and trunk. A series of cameras and computers are used to record the leg position and the walking speed. This data will be compared to the data provided from the device.

DETAILED DESCRIPTION:
This is a comparative cohort study testing the accuracy of a wearable Neural Sleeve in collecting kinematic data in children (age 8-14 years) with CP and healthy control subjects as well as the Sleeve's ability to normalize gait patterns in patients with CP. The Cionic Neural Sleeve measures information on how people move. The system consists of 4 leg straps, 2 foot sensors, and 2 foot insoles (or pressure sensors), connected by insulated wires to a battery-powered control box worn on the thigh. The Cionic sensing devices are made up of sensors that are either part of wearable garments held snugly in place with Velcro and sticky electrode gel, or attached to the shoes. This system will measure and record electromyographic data from the muscles as well as kinematic data in the lower extremities during normal walking speeds in all participants.

All subjects will be examined by a licensed physician or physical therapist prior to fitting the Neural Sleeve. This will consist of lower extremity range of motion, strength testing and selective motor control (all components are part of a typical pediatric orthopaedic neuromuscular physical exam). Thereafter, each participant will be fit for the components of the Cionic Neural Sleeve. Two stretchy leg straps containing multiple sensors will be secured to each leg with Velcro. One strap will be secured around each thigh and one around each shank (lower leg). These straps will measure two things: (1) the activity levels of the muscles underneath the straps, and (2) the physical orientation of the legs. One additional foot sensor will also be attached to the top of each shoe to measure the physical orientation of the subjects feet. The straps and foot sensors will be connected by stretchable wires. Last, thin pressure-sensing pressure pads will be inserted inside each shoe underneath your regular shoe insoles (which will be temporarily removed). The pressure sensors measure where the foot is applying downward pressure inside the shoes at all times. All wires/outputs from sensors will be connected to a battery-powered control box worn at the hip, capable of stimulating muscle contractions (manually or algorithmically). These devices connect wirelessly via Bluetooth to an application running on a smartphone utilized only in the laboratory. The smartphone's camera will record video of the lower body. We will not record the face.

The sleeve will be calibrated through completing a series of tasks while wearing the sleeve for up to 5 minutes, including dorsiflexion/plantarflexion, knee extension and knee flexion. Thereafter, subjects will be asked to then walk at their preferred speed for 2 minutes while the Neural Sleeve collects data only.

Next, all patients will complete a limited instrumented gait analysis. Gait analysis involves recording movement patterns during walking using small reflective markers and sensor taped to the limbs of the subjects. A series of cameras and computers are used to record the kinematic output and temporospatial parameters (speed, cadence, stride width, stride length). Kinematic data from the instrumented gait analysis will be compared to kinematic data collected from the Cionic Neural Sleeve.

Last, in the CP cohort, subjects will be fit with a Functional Electrical Stimulation (FES) control box clipped to the hip or thigh and a maximum of eight pairs (16 total) of sticky electrode pads worn on the shins, calves, quadriceps, and/or hamstrings. These electrodes will connect to the FES control box via insulated wires. FES will then be calibrated to the subject. While seated or lying down, subjects will move their legs and experience targeted FES. FES applies small electrical charges to stimulate the muscle to perform the usual movement, similar to an over-the-counter TENs unit.This will be repeated on each of the 4 main muscle groups: quadriceps, hamstrings, calf, and tibialis anterior (front of lower leg). Each stimulation will last approximately 1 minute long and there will be as much time for rest between stimulations as needed.

CP subjects will then be asked to walk at their preferred speed for up to 2 minutes while the previously-collected EMG data will be used to inform the FES assistance. Kinematic data from collected from the Cionic Neural Sleeve on recording mode only will be compared to FES-assisted kinematic data from the sleeve and from formal gait analysis. They will be sent home with the sleeve to allow for a continuation of the aforementioned analyses over a 12-week period. PROMIS scores will then be collected.

---

sleeve settings: Frequency: 5 Hz to 125 0Hz (5 Hz increments) Pulse width: 100 µs to 400µs (100 µs increments) Intensity: 0 mA to 100 mA (5 mA increments)

A member of the Cionic team will facilitate the configuration and protocol/parameters for the first 2-3 patients while concurrently training members of the study staff. The trained staff member(s) will then take over with device configuration for subsequent patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8-14 years
2. Diagnosis of spastic cerebral palsy affecting one or both legs
3. Able to independently sit, stand and walk with or without assistive device or bracing
4. Able to walk at least 50 feet with or without assistive device or bracing
5. Able to understand and follow basic instructions in English
6. A Parent/Guardian must accompany and be present with the child participant

Exclusion Criteria:

1. Cognitive impairment that would preclude participation
2. Lower motor neuron disease or injury that may impair response to stimulation
3. Diagnosis of any neurologic disease aside from spastic cerebral palsy
4. Dyskinetic movement disorder
5. Have skin conditions of the affected lower limb, including cuts, burns or lesions that would preclude placement of electrodes
6. Have a latex allergy

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Range of motion (degrees) in lower extremities | 2 to 4 hours for formal gait analysis visit
  Participants will be evaluated on range of motion in degrees by performing dorsiflexion, plantarflexion, knee extension, and knee flexion exercises. The physical orientation of both legs and feet, selective motor control, and lower extremity strength will also be evaluated while participants walk for up to two minutes. Specific measures include ambulation speed (km per hour), walking cadence (steps per minute), stride width (inches), and stride length (inches).
  Baseline measures will be obtained in a standard neuromuscular physical exam performed by a licensed physician or physical therapist. During the intervention phase of the study, these measures will be obtained in a formal limited instrument gait analysis while wearing a neural sleeve. Movement patterns will be captured using small reflective markers and sensors to record kinematic output.
Neuromodulation activity (motor unit potential) | 2 to 4 hours for formal gait analysis visit, data collection continuously for 12 weeks after study visit
  Kinematic data from the instrumented gait analysis will be compared to kinematic data collected from the Cionic Neural Sleeve. Specifically, electrical activity, measured by motor unit potential (E-MUP) waveforms and their magnitudes, obtained via electromyography during the gait analysis will be compared to the electrical activity obtained from neuromodulation via the neural sleeve. Neuromodulation will be assessed on the four main muscle groups: quadriceps, hamstrings, calf, and tibialis anterior.

SECONDARY OUTCOMES:
Patient-reported physical function (PROMIS score) | 1 to 2 hours for follow-up clinical visit
  Patient-Reported Outcomes Measurement Information System (PROMIS) scores will be collected from cerebral palsy patients at the conclusion of the 12-week neural sleeve data collection period. The PROMIS questionnaire will generate patient-reported scores to measure physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Thompson, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California - Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data and gait analytics of individual participants with other researchers will not be shared at this time. De-identified IPD may be shared in the future.